CLINICAL TRIAL: NCT01430494
Title: A Multi-center, Longitudinal, Observational Study of Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD) to Establish the Rate, Characteristics, and Determinants of Disease Progression
Brief Title: Observational Study in Patients With Autosomal Dominant Polycystic Kidney Disease
Acronym: OVERTURE
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-10-291
Record Dates: First submitted 2011-07-29; First posted 2011-09-08 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
To collect characteristics of patients with ADPKD across a broad population, over time to better understand disease progression (signs, symptoms and outcomes). Association with total kidney volume changes and other measures of disease progression will be determined in order to identify a population at increased risk for disease progression. The economic and quality life impact of ADPKD will be assessed. Subjects who terminated participation early from clinical trials with tolvaptan may also be followed.

ELIGIBILITY:
Inclusion Criteria:

* existing diagnosis of ADPKD by modified-Ravine criteria
* Total kidney volume >= 300 cc/m height by ultrasound or >= 250 cc/m height by MRI

Exclusion Criteria:

* Current or expected (within the next six months) interventions for the treatment of ADPKD affecting kidney volume

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be identified by participating clinics (primarily nephrology clinics) treating patients with ADPKD.
Sampling Method: Non-Probability Sample
Enrollment: 3409 (Actual)
Dates: Start 2011-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Correlation of change in total kidney volume with ADPKD-related outcomes | 1 year

SECONDARY OUTCOMES:
Patient-reported pain | every 6 months
SF-12 Scores | every 6 months
ADPKD-Impact Scale Score | every 6 months
Cost of care | every 6 months
EQ-5D Scores | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Czerwiec, MD, PhD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (234):
- United States (93):
  - Otsuka Investigational Site 1, Peoria, Arizona
  - Otsuka Investigational Site 2, Peoria, Arizona
  - Otsuka Investigational Site, Tempe, Arizona
  - Otsuka Investigational Site, Azusa, California
  - Otsuka Investigational Site, Bakersfield, California
  - Otsuka Investigational Site, Los Angeles, California
  - Otsuka Investigational Site, Ontario, California
  - Otsuka Investigational Site, San Diego, California
  - Otsuka Investigational Site, Arvada, Colorado
  - Otsuka Investigational Site, Aurora, Colorado
  - Otsuka Investigational Site, Denver, Colorado
  - Otsuka Investigational Site, New Haven, Connecticut
  - Otsuka Investigational Site, Washington D.C., District of Columbia
  - Otsuka Investigational Site, Coral Gables, Florida
  - Otsuka Investigational Site, Hudson, Florida
  - Otsuka Investigational Site, Jacksonville, Florida
  - Otsuka Investigational Site, Melbourne, Florida
  - Otsuka Investigational Site, Port Charlotte, Florida
  - Otsuka Investigational Site, Tampa, Florida
  - Otsuka Investigational Site, Atlanta, Georgia
  - Otsuka Investigational Site, Augusta, Georgia
  - Otsuka Investigational Site, Meridian, Idaho
  - Otsuka Investigational Site, Chicago, Illinois
  - Otsuka Investigational Site, Peoria, Illinois
  - Otsuka Investigational Site, Mishawaka, Indiana
  - Otsuka Investigational Site, Kansas City, Kansas
  - Otsuka Investigational Site, Wichita, Kansas
  - Otsuka Investigational Site, Lexington, Kentucky
  - Otsuka Investigational Site, Paducah, Kentucky
  - Otsuka Investigational Site, New Orleans, Louisiana
  - Otsuka Investigational Site, Baltimore, Maryland
  - Otsuka Investigational Site, Bethesda, Maryland
  - Otsuka Investigational Site, Rockville, Maryland
  - Otsuka Investigational Site, Wheaton, Maryland
  - Otsuka Investigational Site, Boston, Massachusetts
  - Otuska Investigational Site, Holyoke, Massachusetts
  - Otsuka Investigational Site, Plymouth, Massachusetts
  - Otsuka Investigational Site, Springfield, Massachusetts
  - Otsuka Investigational Site, Detroit, Michigan
  - Otsuka Investigational Site, Kalamazoo, Michigan
  - Otsuka Investigational Site, Pontiac, Michigan
  - Otsuka Investigational Site, Royal Oak, Michigan
  - Otsuka Investigational Site, Brooklyn Center, Minnesota
  - Otsuka Investigational Site, Rochester, Minnesota
  - Otsuka Investigational Site, St Louis, Missouri
  - Otsuka Investigational Site, Las Vegas, Nevada
  - Otsuka Investigational Site, Reno, Nevada
  - Otsuka Investigational Site, Mount Laurel, New Jersey
  - Otsuka Investigational Site, Princeton Junction, New Jersey
  - Otsuka Investigational Site, Voorhees Township, New Jersey
  - Otsuka Investigational Site, Albuquerque, New Mexico
  - Otsuka Investigational Site, Albany, New York
  - Otsuka Investigational Site, Brooklyn, New York
  - Otsuka Investigational Site, Buffalo, New York
  - Otsuka Investigational Site, Flushing, New York
  - Otsuka Investigational Site, Forest Hills, New York
  - Otsuka Investigational Site, Great Neck, New York
  - Otsuka Investigational Site, Mineola, New York
  - Otsuka Investigational Site, New York, New York
  - Otsuka Investigational Site, Port Washington, New York
  - Otsuka Investigational Site, Rochester, New York
  - Otsuka Investigational Site, Rosedale, New York
  - Otsuka Investigational Site, The Bronx, New York
  - Otsuka Investigational Site, Chapel Hill, North Carolina
  - Otsuka Investigational Site, Durham, North Carolina
  - Otsuka Investigational Site, Winston-Salem, North Carolina
  - Otsuka Investigational Site, Devils Lake, North Dakota
  - Otsuka Investigational Site, Fargo, North Dakota
  - Otsuka Investigational Site, Cincinnati, Ohio
  - Otsuka Investigational Site, Cleveland, Ohio
  - Otsuka Investigational Site, Columbus, Ohio
  - Otsuka Investigational Site, Portland, Oregon
  - Otsuka Investigational Site, Altoona, Pennsylvania
  - Otsuka Investigational Site, Bethleham, Pennsylvania
  - Otsuka Investigational Site, Doylestown, Pennsylvania
  - Otsuka Investigational Site, Lancaster, Pennsylvania
  - Otsuka Investigational Site, Philadelphia, Pennsylvania
  - Otsuka Investigational Site, Providence, Rhode Island
  - Otsuka Investigational Site, Aiken, South Carolina
  - Otsuka Investigational Site, Anderson, South Carolina
  - Otsuka Investigational Site, Columbia, South Carolina
  - Otsuka Investigational Site, Rapid City, South Dakota
  - Otsuka Investigational Site, Knoxville, Tennessee
  - Otsuka Investigational Site, Arlington, Texas
  - Otsuka Investigational Site, Fort Worth, Texas
  - Otsuka Investigational Site, Houston, Texas
  - Otsuka Investigational Site, Mission, Texas
  - Otsuka Investigational Site, San Antonio, Texas
  - Otsuka Investigational Site, Burlington, Vermont
  - Otsuka Investigational Site, Fairfax, Virginia
  - Otsuka Investigational Site, Bluefield, West Virginia
  - Otsuka Investigational Site, Morgantown, West Virginia
  - Otsuka Investigational Site, Madison, Wisconsin
- Argentina (11):
  - Otsuka Investigational Site, Avellaneda, Buenos Aires
  - Otsuka Investigational Site, Junín, Buenos Aires
  - Otsuka Investigational Site, La Plata, Buenos Aires
  - Otsuka Investigational Sites, Pergamino, Buenos Aires
  - Otsuka Investigational Site, Pilar, Buenos Aires
  - Otsuka Investigational Site, Buenos Aires, C.a.b.a.
  - Otsuka Investigational Site, Córdoba, Córdoba Province
  - Otsuka Investigational Site, Buenos Aires
  - Otsuka Investigational Site, Ciudad de Buenos Aires
  - Otsuka Investigational Site, Córdoba
  - Otsuka Investigational Site, Sante Fe
- Australia (11):
  - Otsuka Investigational Site, Liverpool, New South Wales
  - Otsuka Investigational Site, Newcastle, New South Wales
  - Otsuka Investigational Site, Sydney, New South Wales
  - Otsuka Investigational Site, Westmead, New South Wales
  - Otsuka Investigational Site, Adelaide, South Australia
  - Otsuka Investigational Site, Launceston, Tasmania
  - Otsuka Investigational Site, Clayton, Victoria
  - Otsuka Investigational Site, Melbourne, Victoria
  - Otsuka Investigational Site, Parkville, Victoria
  - Otsuka Investigational Site, Richmond, Victoria
  - Otsuka Investigational Site, Perth, Western Australia
- Belgium (3):
  - Otsuka Investigational Site, Brussels
  - Otsuka Investigational Site, Ghent
  - Otsuka Investigational Site, Leuven
- Brazil (7):
  - Otsuka Investigational Site, Belo Horizonte, Minas Gerais
  - Otsuka Investigational Site, Juiz de Fora, Minas Gerais
  - Otsuka Investigational Site, Curitiba, Paraná
  - Otsuka Investigational Site, Porto Alegre, Rio Grande do Sul
  - Otsuka Investigational Site, Joinville, Santa Catarina
  - Otsuka Investigational Site, São José do Rio Preto, São Paulo
  - Otsuka Investigational Site, São Paulo, São Paulo
- Canada (10):
  - Otsuka Investigational Site, Vancouver, British Columbia
  - Otsuka Investigational Site, St. John's, Newfoundland and Labrador
  - Otsuka Investigational Site, Halifax, Nova Scotia
  - Otsuka Investigational Site, Brampton, Ontario
  - Otsuka Investigational Site, Edmonton, Ontario
  - Otsuka Investigational Site, Oakville, Ontario
  - Otsuka Investigational Site, Scarborough Village, Ontario
  - Otsuka Investigational Site, Toronto, Ontario
  - Otsuka Investigational Site, Greenfield Park, Quebec
  - Otsuka Investigational Site, Montreal, Quebec
- Czechia (5):
  - Otsuka Investigational Site, České Budějovice
  - Otsuka Investigational Site, Hradec Králové
  - Otsuka Investigational Site, Jihlava
  - Otsuka Investigational Site, Liberec
  - Otsuka Investigational Site, Prague
- France (7):
  - Otsuka Investigational Site, Caen
  - Otsuka Investigational Site, Grenoble
  - Otuska Investigational Site, Lyon
  - Otsuka Investigational Site, Lyon
  - Otsuka Investigational Site, Montpellier
  - Otsuka Investigational Site, Pierre-Bénite
  - Otsuka Investigational Site, Vandœuvre-lès-Nancy
- Germany (8):
  - Otsuka Investigational Site, Berlin
  - Otsuka Investigational Site, Dresden
  - Otsuka Investigational Site, Düsseldorf
  - Otsuka Investigational Site, Erlangen
  - Otsuka Investigational Site, Hanover
  - Otsuka Investigational Site, Heidelberg
  - Otsuka Investigational Site, Munich
  - Otsuka Investigational Site, Wiesbaden
- Italy (7):
  - Otsuka Investigational Site, Rozzano, Milano
  - Otsuka Investigational Site, Bologna
  - Otsuka Investigational Site, Lecco
  - Otsuka Investigational Site, Modena
  - Otsuka Investigational Site, Montichiari, (Brescia)
  - Otsuka Investigational Site, Napoli
  - Otsuka Investigational Site, Pavia
- Japan (9):
  - Otsuka Investigational Site, Sagamihara-shi, Kanagawa
  - Otsuka Investigational Site, Kurashiki, Okayama-ken
  - Otsuka Investigational Site, Chiba
  - Otsuka Investigational Site, Fukuoka
  - Otsuka Investigational Site, Hokkaido
  - Otsuka Investigational Site, Niigata
  - Otsuka Investigational Site, Osaka
  - Otsuka Investigational Site, Tochigi
  - Otsuka Investigational Site, Tokyo
- Netherlands (4):
  - Otsuka Investigational Site, Groningen
  - Otsuka Investigational Site, Leiden
  - Otsuka Investigational Site, Nijmegen
  - Otsuka Investigational Site, Rotterdam
- Norway (2):
  - Otsuka Investigational Site, Drammen
  - Otsuka Investigational Site, Lillehammer
- Poland (9):
  - Otsuka Investigational Site, Ciechanów
  - Otsuka Investigational Site, Golub-Dobrzyń
  - Otsuka Investigational Site, Krakow
  - Otsuka Investigational Site, Lodz
  - Otsuka Investigational Site, Radom
  - Otsuka Investigational Site, Rzeszów
  - Otsuka Investigational Site, Szczecin
  - Otsuka Investigational Site, Warsaw
  - Otsuka Investigational Site, Wroclaw
- Romania (3):
  - Otsuka Investigational Site, Oradea, Bihor County
  - Otsuka Investigational Site, Timișoara, Timiș County
  - Otsuka Investigational Site, Bucharest
- Spain (5):
  - Otsuka Investigational Site, Alicante
  - Otsuka Investigational Site, Barcelona
  - Otsuka Investigational Site, Ciudad Real
  - Otsuka Investigational Site, Hospitalet de Ilobre
  - Otsuka Investigational Site, Madrid
- Sweden (2):
  - Otsuka Investigational Site, Malmo
  - Otsuka Investigational Site, Stockholm
- Otsuka Investigational Site, Zurich, Switzerland
- Turkey (Türkiye) (6):
  - Otsuka Investigational Site, Istanbul, Capa
  - Otsuka Investigational Site, Inciraltı, İzmir
  - Otsuka Investigational Site, Balcali-Adana
  - Otsuka Investigational Site, Bornova-Izmir
  - Otsuka Investigational Site, Izmir
  - Otsuka Investigational Site, Sihhiye-Ankara
- United Kingdom (31):
  - Otsuka Investigational Site, Exeter, Devon
  - Otsuka Investigational Site, York, North Yorkshire
  - Otsuka Investigational Site, Stoke-on-Trent, Staffordshire
  - Otsuka Investigational Site, Carshalton, Surrey
  - Otsuka Investigational Site, Birmingham, West Midlands
  - Otsuka Investigational Site, Belfast
  - Otsuka Investigational Site, Bradford
  - Otsuka Investigational Site, Bristol
  - Otsuka Investigational Site, Cambridge
  - Otsuka Investigational Site, Chelmsford
  - Otsuka Investigational Site, Coventry
  - Otsuka Investigational Site, Dorchester
  - Otsuka Investigational Site, Edinburgh
  - Otsuka Investigational Site, Hull
  - Otsuka Investigational Site, Inverness
  - Otsuka Investigational Site, Kirkcaldy
  - Otsuka Investigational Site, Leicester
  - Otsuka Investigational Site, Liverpool
  - Otsuka Investigational Site, London
  - Otsuka Investigational Site, Manchester
  - Otsuka Investigational Site, Middlesbrough
  - Otsuka Investigational Site, Newcastle upon Tyne
  - Otsuka Investigational Site, Oxford
  - Otsuka Investigational Site, Portsmouth
  - Otsuka Investigational Site, Preston
  - Otsuka Investigational Site, Salford
  - Otsuka Investigational Site, Sheffield
  - Otsuka Investigational Site, Southampton
  - Otsuka Investigational Site, Stevenage
  - Otsuka Investigational Site, Westcliff-on-Sea
  - Otsuka Investigational Site, Wolverhampton

REFERENCES:
- [Derived] Gitomer BY, Chonchol M, Zhou X, Garbinsky D, Wang J, Nunna S, Fernandes AW, Oberdhan D. Kidney Stone Disease and Progression Risk in Autosomal Dominant Polycystic Kidney Disease: A Post Hoc Analysis of OVERTURE. Kidney360. 2024 Sep 1;5(9):1364-1366. doi: 10.34067/KID.0000000000000524. Epub 2024 Jul 24. No abstract available. PMID 39752236
- [Derived] Lioudis M, Zhou X, Davenport E, Nunna S, Krasa HB, Oberdhan D, Fernandes AW. Effects of tolvaptan discontinuation in patients with autosomal dominant polycystic kidney disease: a post hoc pooled analysis. BMC Nephrol. 2023 Jun 22;24(1):182. doi: 10.1186/s12882-023-03247-6. PMID 37349694
- [Derived] Chebib FT, Zhou X, Garbinsky D, Davenport E, Nunna S, Oberdhan D, Fernandes A. Tolvaptan and Kidney Function Decline in Older Individuals With Autosomal Dominant Polycystic Kidney Disease: A Pooled Analysis of Randomized Clinical Trials and Observational Studies. Kidney Med. 2023 Apr 14;5(6):100639. doi: 10.1016/j.xkme.2023.100639. eCollection 2023 Jun. PMID 37250503
- [Derived] Perrone RD, Oberdhan D, Ouyang J, Bichet DG, Budde K, Chapman AB, Gitomer BY, Horie S, Ong ACM, Torres VE, Turner AN, Krasa H. OVERTURE: A Worldwide, Prospective, Observational Study of Disease Characteristics in Patients With ADPKD. Kidney Int Rep. 2023 Feb 13;8(5):989-1001. doi: 10.1016/j.ekir.2023.02.1073. eCollection 2023 May. PMID 37180499